CLINICAL TRIAL: NCT03830242
Title: Diagnostic Significance of Single Center, Open and Prospective Evaluation of <Sup>18<Sup>F-FDG PET/CT Dynamic Imaging in Detecting Metastatic Central Lymph Nodes in Patients With Papillary Thyroid Cancer
Brief Title: Diagnostic Significance of FDG PET/CT Dynamic Imaging in Detecting Metastatic Lymph Nodes With Papillary Thyroid Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hongjun Jin, principal Investigator, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ZDWY.JRWK.001
Record Dates: First submitted 2018-12-17; First posted 2019-02-05 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Positron-Emission Tomography; Lymph Node Metastases; Thyroid Cancer
MeSH Terms: conditions — Lymphatic Metastasis; Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- <Sup>18<Sup>F-FDG PET/CT study group (Experimental): <Sup>18<Sup>F-FDG PET/CT dynamic scan,Pathological examination and gene detection Diagnostic Test: <Sup>18<Sup>F-FDG PET/CT dynamic scan The purpose of this study is to carry out <Sup>18<Sup>F-FDG PET/CT dynamic scans and Pathological examination of metastatic central lymph nodes in newly diagnosed patients with papillary thyroid cancer, and to compare imaging findings, genomics, and pathology at the same time. The intrinsic relationship between tissue characteristics and the diagnostic value of <Sup>18<Sup>F-FDG PET/CT dynamic imaging in metastatic central lymph nodes with papillary thyroid cancer are discussed.
  Interventions: Diagnostic Test: <Sup>18<Sup>F-FDG PET/CT dynamic scan
- B-ultrasonography group (Other): B-ultrasonography,Pathological examination and gene detection Diagnostic Test:B-ultrasonography The purpose of this study is to carry out <Sup>18<Sup>F-FDG PET/CT dynamic scans and Pathological examination of metastatic central lymph nodes in newly diagnosed patients with papillary thyroid cancer, and to compare imaging findings of B-ultrasonography , genomics, and pathology at the same time. The intrinsic relationship between tissue characteristics and the diagnostic value of <Sup>18<Sup>F-FDG PET/CT dynamic imaging in metastatic central lymph nodes with papillary thyroid cancer are discussed.
  Interventions: Diagnostic Test: B-ultrasonography

INTERVENTIONS:
Diagnostic Test: <Sup>18<Sup>F-FDG PET/CT dynamic scan — The purpose of this study is to carry out <Sup>18<Sup>F-FDG PET/CT dynamic scans and Pathological examination of metastatic central lymph nodes in newly diagnosed patients with papillary thyroid cancer, and to compare imaging findings, genomics, and pathology at the same time. The intrinsic relationship between tissue characteristics and the diagnostic value of <Sup>18<Sup>F-FDG PET/CT dynamic imaging in metastatic central lymph nodes with papillary thyroid cancer are discussed.
  Arms: <Sup>18<Sup>F-FDG PET/CT study group
Diagnostic Test: B-ultrasonography — The purpose of this study is to carry out <Sup>18<Sup>F-FDG PET/CT dynamic scans and Pathological examination of metastatic central lymph nodes in newly diagnosed patients with papillary thyroid cancer, and to compare imaging findings of B-ultrasonography , genomics, and pathology at the same time. The intrinsic relationship between tissue characteristics and the diagnostic value of <Sup>18<Sup>F-FDG PET/CT dynamic imaging in metastatic central lymph nodes with papillary thyroid cancer are discussed.
  Arms: B-ultrasonography group

SUMMARY:
The aim of this study is to make up for the gap by performing a dynamic scan of <Sup>18<Sup>F-FDG PET/CT on newly diagnosed patients with papillary thyroid carcinoma. Pathological and genomic studies are performed. The differences between metastatic central lymph nodes images and tissues are compared at the same time. <Sup>18<Sup>F-FDG PET/CT dynamic imaging is explored in metastatic central lymph nodes with papillary thyroid cancer for the diagnostic value.

DETAILED DESCRIPTION:
Thyroid cancer is the most common malignant tumor in human endocrine system, accounting for 0.2% ~ 1.0% of malignant tumors .According to the global cancer report released by the world health organization (WHO) in 2014, 50% of the new cases of thyroid cancer are papillary thyroid cancer (PTC). In recent years, the incidence of thyroid cancer in China shows an increasing trend, especially the composition ratio of thyroid micro-papillary carcinoma with the focal diameter <1 cm increases rapidly.Although PTC has a good prognosis, according to a Meta analysis , PTC lymph node metastasis rate is as high as 28.0%.The central lymph node is the most common metastatic site of papillary thyroid carcinoma.In addition, it has been reported in literature that lymph nodes in the central region are the first stop of thyroid papillary carcinoma metastasis (i.e., sentinel lymph nodes), and lymph nodes metastatic to this point are prone to infringe the peripheral esophagus, trachea and recurrent laryngeal nerve at an early stage.A large number of clinical cases have confirmed that lymph node metastasis of thyroid cancer significantly increases the local recurrence rate after surgery.More studies have shown that regional lymph node metastasis increases mortality.Therefore, the treatment of lymph node metastasis should not be ignored in PTC patients.However, at present, preoperative imaging has certain limitations in the judgment of lymph node metastasis in the central region : ultrasound has advantages in the judgment of lymph node metastasis in the peripheral group, but poor display in the central group.Although MRI scan of head and neck can be multi-directional and multi-sequence imaging, and the resolution of soft tissue is high, it is not good at showing calcification.Conventional CT alone based on lymph node morphology to determine metastasis also has some limitations;Positron emission tomography (PET) sensitivity was < 40%.Although one study showed that the probability of non-missed diagnosis of lymph nodes in central PTC region by thin slice CT scan was 100%, the specificity was low and the study was retrospective.Therefore, b-ultrasound, MRI, CT, PET and other auxiliary examinations have not been able to effectively detect all central metastatic lymph nodes before surgery.For management of cervical lymph nodes ,2015 American Thyroid Association（ATA） guidelines show that thyroid+therapeutic Ⅵ area lymph node dissection should be undertaken if in central or lateral lymph nodes are involved.Chinese guidelines recommend that, in order to avoid operative complications as far as possible (i.e. effective retainment of the parathyroid gland and recurrent laryngeal nerve), regardless of the size of the primary thyroid lesion, lymph node dissection in the central area on the same side of the lesion should be performed at least.However, in 2017, the second edition of National Comprehensive Cancer Network(NCCN) thyroid tumor guidelines believed that if lymph nodes in the central region were negative, preventive central region lymph node dissection was not recommended.Above all，there is so much controversy over lymph node dissection in the central region. Therefore，it is of great significance to effectively evaluate the preoperative lymph nodes station in the central region of thyroid papillary carcinoma.

Early dynamic imaging examination of <Sup>18<Sup>F-FDG PET/CT can be defined as a imaging method to detect the status of radioactive tracer (<Sup>18<Sup>F-FDG) which travels with the blood flow and is continuously absorbed and excreted by organs (or diseased) tissues after being introduced into the body in the early stage.This development reflects the change of <Sup>18<Sup>F-FDG activity with time in the early stage of entering the body, and can provide information about the dynamic change of tracer metabolism and distribution in tissues with time, so that it can provide more metabolic and distribution details of tumor lesions and metastatic lesions than static scanning.At present, many studies have shown that <Sup>18<Sup>F-FDG PET/CT early dynamic imaging technology can effectively improve the sensitivity of hepatocellular carcinoma ,renal cell carcinoma and other tumors.More amazing，there may be more advantages in evaluating lymph node metastasis.The blood supply of lymph nodes metastatic of thyroid papillary carcinoma is abundant, which helps to locate the metastatic tumor lymph node.However，there is no relevant study.Now , investigators plan to observe the significance of the method to evaluate the central lymph node metastasis in thyroid papillary carcinoma as well as the intrinsic correlations between the significance and postoperative pathological results ,which may help to develop surgical strategy by preoperative evaluation and avoiding additional dissection.

ELIGIBILITY:
Inclusion Criteria:

* • Accurately diagnosing primary papillary thyroid cancer according to pathological diagnostic criteria .

  * Thyroid papillary carcinoma was suspected by thyroid ultrasound text and/or neck CT.
  * The age is more than 18 years old and less than 65 years old. There is no gender restriction.
  * Untreated patients who have not received surgery, interventional therapy,chemotherapy, biotherapy, and radiation therapy.
  * Physical condition score of Eastern Cooperative Oncology Group（ECOG）: 0-2; no major organ dysfunction; oxygen partial pressure ≥ 10.64 kilopascal（kPa）; white blood cell count≥ 4 × 109/L; hemoglobin≥ 9.5g/dL; neutrophil absolute count ≥ 1.5 × 109 / L; platelet count ≥ 100× 109 / L; total bilirubin ≤ 1.5 times of the upper limit of normal value;creatinine ≤ 1.25 times of the upper limit of normal value; and creatinine clearance ≥ 60ml / min.
  * Be able to obtain complete follow-up information, understand the situation of this study and sign informed consent.

Exclusion Criteria:

* • Poorly controlled diabetics (fasting blood glucose levels > 200 mg/dL).• In addition to four types of malignant tumors that can be treated with radical resection, such as cervical cancer in situ, basal or squamous cell skin cancer, (breast) ductal carcinoma in situ, and organ localized prostate cancer, suffering from any other malignant tumors within 5 years.• Breastfeeding and/or pregnant women.

  * Patients with severe bleeding tendencies (prothrombin time less than 50%,cannot be corrected by treatment with vitamin K, etc.).
  * Recent severe hemoptysis, severe cough, dyspnea or patients are not able to cooperate.
  * People with severe emphysema, pulmonary congestion, and pulmonary heart disease.
  * Researchers believe that the subject may not be able to complete this study or may not be able to comply with the requirements of this study (for management reasons or other reasons).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of lymph nodes dissected | 12 months
  Count the number of lymph nodes dissected during operation of every Participants.
Number of Participants diagnosed with lymph node metastasis by <Sup>18<Sup>F-FDG PET/CT dynamic scans. | 12 months
  Count the number of Participants diagnosed with lymph node metastasis by <Sup>18<Sup>F-FDG PET/CT dynamic scans.
Number of Participants diagnosed with lymph node metastasis by Postoperative pathology | 12 months
  Count the number of Participants diagnosed with lymph node metastasis by Postoperative pathology.
The number of lymph node metastases in patients with different Genetic types | 12 months
  To count the number of lymph node metastases in patients with different Genetic types basing on genetic testing.

SECONDARY OUTCOMES:
Calculating the overall diagnostic sensitivity of <Sup>18<Sup>F-FDG PET/CT dynamic scans | 12 months
  Calculating the overall diagnostic sensitivity based on the results of <Sup>18<Sup>F-FDG PET/CT dynamic scans and Postoperative pathology.
Calculating the overall diagnostic specificity of <Sup>18<Sup>F-FDG PET/CT dynamic scans | 12 months
  Calculating the overall diagnostic specificity based on the results of <Sup>18<Sup>F-FDG PET/CT dynamic scans and Postoperative pathology.
Calculating the receiver operating characteristic curve（ROC） | 12 months
  Calculate receiver operating characteristic curve（ROC） based on sensitivity and specificity.
Calculating the radionics indicators of <Sup>18<Sup>F-FDG PET/CT | 12 months
  Based on the results above,to calculate the radionics indicators of <Sup>18<Sup>F-FDG PET/CT dynamic scans in detecting metastatic central lymph nodes in participants with papillary thyroid cancer .

CONTACTS AND LOCATIONS:
Locations (1):
- Fifth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided